CLINICAL TRIAL: NCT07133854
Title: The Impact of Adipose Tissue Insulin Resistance and Abdominal Obesity on Hepatic Fatty Acid Metabolism in Type 1 Diabetes
Brief Title: How Abnormal Function of Fat Tissue in Type 1 Diabetes Contributes to Fat in the Liver
Acronym: AGL14
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenure professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2026-5900
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Non-Alcoholic Steato-Hepatitis (NASH); Type 1 Diabetes Mellitus
Keywords: abdominal obesity; Adipose tissue insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with Type 1 Diabetes (Experimental): Participants will undergo a 9-hour postprandial metabolic study
  Interventions: Diagnostic Test: Imaging PET/MRI; Diagnostic Test: Stable isotope infusions; Diagnostic Test: meal test; Diagnostic Test: Indirect calorimetry
- Group without Type 1 Diabetes (Experimental): Participants will undergo a 9-hour postprandial metabolic study
  Interventions: Diagnostic Test: Imaging PET/MRI; Diagnostic Test: Stable isotope infusions; Diagnostic Test: meal test; Diagnostic Test: Indirect calorimetry

INTERVENTIONS:
Diagnostic Test: Imaging PET/MRI — MRI using 1H-MRS and Dixon sequences on a 3 T clinical MRI system (Ingenia, Philips Healthcare, Best, the Netherlands) will be performed.
  [11C]-palmitate: 1 x i.v. injection of 175 MBq followed by TEP imaging. [18F]-FTHA: oral administration of 75 MBq followed by TEP imaging.
Diagnostic Test: Stable isotope infusions — [6,6 D2]-glucose infusion (0.22 µmol/kg/min, preceded by a bolus of 22 µmol/kg) will start from -180 until time + 360.
  [1,1,2,3,3-2H]-glycerol (0.05 µmol/kg/min.) and of [7,7,8,8-2H] palmitate (0.01 µmol/kg/min) will start from time -60 until time +360.
Diagnostic Test: meal test — A liquid meal will be administered at time 0. The liquid meal (400 ml) energy breakdown is 50% (101g) from glucose, 33% (31g) from fat, and 17% (40g) from protein; participants will consume the 400 ml in 4 aliquots of 100 ml over 20 min, supplemented with 0.9 g of U-[13C]-glucose and 9 μmol/kg lean mass of [U-13C]-palmitate.
Diagnostic Test: Indirect calorimetry — Indirect calorimetry (Vmax Series from Vyaire medical, licence # 22536), measured during10 minutes, every hour.

SUMMARY:
Steatotic liver disease associated with metabolic dysfunction (MASLD) is a disease caused by excess fat storage in the liver. Excessive fat delivery to the liver and MASLD typically occurs in people with abdominal obesity and type 2 diabetes. Type 1 diabetes (T1D) is also associated with a marked increase in the release of fat from adipose tissues and MASLD is increased in T1D and significantly increases the risk of heart, kidney and eye diseases.

DETAILED DESCRIPTION:
It is a parallel study design between T1D and controls. The outcomes will be assessed between T1D vs. controls during the metabolic visit.

The metabolic visit will last 9 hours: it will be a test meal with perfusion of stable tracers, blood sampling, PET acquisitions using radiopharmaceuticals (18FTHA and 11C-palmitate) and MRI acquisitions.

In total, 32 participants will be recruited:

* 16 living with T1D and abdominal obesity
* 16 with normoglycemia

ELIGIBILITY:
Inclusion Criteria:

* 16 individuals living with T1D and abdominal obesity, as defined by the International Diabetes Federation country/ethnic group-specific criteria (https://www.idf.org/e-library/consensus-statements/60- [1]. Treatment for T1D will be intensive insulin therapy on continuous pump perfusion with continuous glucose monitoring.
* 16 individuals with normoglycemia (i.e., HbA1c below 6.0%) matched for sex, age (± 5 years), waist circumference (± 3 cm), and menopausal status.

Exclusion Criteria:

* less than 70% of time in glycemic range (for T1D);
* history of primary dyslipidemia (LDL-cholesterol over 5 mmol/L or TG over 10 mmol/L) or uncontrolled high blood pressure (over 160/100 mmHg) precluding the withdrawal of lipid lowering and anti-hypertensive agents as per protocol;
* presence of overt cardiovascular, liver or renal disease (except microalbuminuria without reduced kidney function), or other uncontrolled medical conditions;
* use of any medication other than insulin that may affect lipid or carbohydrate metabolism and that cannot be stopped prior to testing;
* current or planned pregnancy within the next 6 months;
* any contraindication to MRI.
* Being allergic to eggs
* Smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day
* Having participated to a research study with exposure to radiation in the last year before the start of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
hepatic NEFA uptake | At baseline of Visit 2 (V2)
  using 11C-palmitate PET

SECONDARY OUTCOMES:
postprandial hepatic Dietary Fatty Acid uptake | At V2 (from time 0 to +360 minutes)
  using 18F-FTHA
Adipose Tissue DFA trapping and postprandial palmitate flux | At V2 (from time 0 to +360 minutes)
  Determined from the same static (whole-body) acquisition image using oral administration of [18F]-Fluoro-6-Thia- Heptadecanoic Acid (FTHA)
hepatic fatty acid oxidation, esterification and secretion into VLDL | At baseline
  [11C]-Palmitate PET. Calculated from the same multicompartmental equation using liver [11C]-palmitate kinetics
Hepatic triglyceride content | At V2 (-200 minutes)
  measured by MRI
Endogenous Glucose production and meal glucose systemic flux | At V2 (from time 0 to +360 minutes)
  Apparition rate (µmol/min) of glucose from multicompartimental equation using intravenous perfusion and oral stable isotope tracer
Insulin secretion | At V2 (from time 0 to +360 minutes)
  Determined by measuring C-peptide kinetics following the liquid meal
Insulin resistance/ sensitivity | At V2 (from time 0 to +360 minutes)
  Determined by measuring circulating glucose and insulin following the liquid meal: glucose and insulin will be combined to give insulin resistance/sensitivity
Glycerol turnover | At visit 2 (from time 0 to +360 minutes)
  calculated from [1,1,2,3,3-2H]-glycerol i.v.
Total substrate utilisation | At visit 2 (from time 0 to +360 minutes).
  measured by using indirect calorimetry
metabolite response | At visit 2 (from time 0 to +360 minutes)
  Colorimetric assay
hormonal response | At visit 2 (from time 0 to +360 minutes)
  Multiplex assay
plasma NEFA NEFA flux | At visit 2 (from time 0 to +360 minutes)
  calculated from i.v. stable isotope tracer (mass spectrometry).
plasma distribution of DFA metabolites | At visit 2 (from time 0 to +360 minutes)
  calculated from i.v. and oral stable isotope tracers (mass spectrometry) incorporated into triglyceride-rich lipoproteins and NEFA.
Adipose tissue Insulin Resistance index | At visit 2 (from time 0 to +360 minutes)
  is calculated from measurement of postabsorptive concentrations of FFAs and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: André C Carpentier, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada